CLINICAL TRIAL: NCT06644625
Title: CHAAMP (CHArlotte Advocate MGUS Project) Internal Pilot Study
Status: Recruiting | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Atrium Health Levine Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00107462; LCI-PCD-MGUS-SCRN-001 (Other: Atrium Health Wake Forest Baptist Comprehensive Cancer Center); NCI-2025-00147 (Other: National Cancer Institute)
Record Dates: First submitted 2024-09-27; First posted 2024-10-16 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma; Multiple Myeloma Progression; Monoclonal Gammopathy of Undetermined Significance (MGUS); Smoldering Multiple Myeloma (SMM); Plasma Cell Disorders
Keywords: multiple myeloma; hematology; plasma cell disorders
MeSH Terms: conditions — Multiple Myeloma; Monoclonal Gammopathy of Undetermined Significance; Smoldering Multiple Myeloma | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and buccal swab
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MGUS and Smoldering Multiple Myeloma: Participants diagnosed with MGUS and smoldering multiple myeloma
  Interventions: Other: Blood draw for the laboratory assessment
- Other Plasma Cell Disorders: Participants diagnosed with other plasma cell disorders
  Interventions: Other: Blood draw for the laboratory assessment

INTERVENTIONS:
Other: Blood draw for the laboratory assessment — Screening blood sample collection to test for MGUS

SUMMARY:
The purpose of this study is to identify multiple myeloma in the precancerous MGUS stage in order to reduce the risk of delayed diagnosis of multiple myeloma, decrease morbidity related to multiple myeloma at progression, and improve long term outcomes.

DETAILED DESCRIPTION:
The CHAAMP Internal Pilot is a pilot and feasibility study conducted to evaluate the feasibility of the trial methods before a full-scale screening effort is launched. High risk individuals 30 years of age or older residing in Charlotte or surrounding area will be screened for MGUS over one-year period with a target enrollment of 1665 participants. Individuals screening positive for monoclonal gammopathy will be provided a clinic referral for further diagnostic evaluation to confirm MGUS, SMM, or other PCD-related disorder, and will be given the opportunity to consent for the Longitudinal portion of the study. Participants diagnosed with MGUS and smoldering multiple myeloma will be prospectively followed for 10 years per protocol. Participants diagnosed with other plasma cell disorders will have their diagnosis and baseline data captured in the registry and followed for overall survival only.

ELIGIBILITY:
SCREENING Inclusion Criteria:

* Age 30 years or older at the time of consent
* Either:

  1. Self-identify as Black and/or African American OR
  2. First-degree relatives (parents, siblings, or children) of patients of any race or ethnicity diagnosed with a plasma cell disorder, including MGUS, smoldering multiple myeloma (SMM), multiple myeloma (MM), solitary plasmacytoma, plasma cell leukemia, AL amyloidosis, POEMS syndrome, and Waldenström's Macroglobulinemia
* Capable and willing to provide informed consent. NOTE: HIPAA (Health Insurance Portability and Accountability Act) authorization for the release of personal health information may be included in the informed consent or obtained separately
* Reside in Charlotte, NC, or the surrounding area, based on self-report

SCREENING Exclusion Criteria:

* Self-reported history of MGUS, SMM, MM, AL amyloidosis, plasma cell leukemia, solitary plasmacytoma, Waldenstrom Macroglobulinemia, and POEMS.

LONGITUDINAL Inclusion Criteria:

* Test positive for monoclonal gammopathy during screening portion of the study
* Consent to the longitudinal portion of the study

LONGITUDINAL Exclusion Criteria:

* The participant previously underwent diagnostic work up as part of CHAAMP Internal Pilot that did not result in a diagnosis of MGUS, Smoldering Multiple Myeloma or other non-plasma cell disorder.

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: High risk individuals with age greater than or equal to 30 years at the time of consent, residing in the Charlotte, NC or surrounding areas.
Sampling Method: Non-Probability Sample
Enrollment: 1665 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2035-01 (Estimated); Study Completion 2035-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants who were Enrolled | Baseline, for an accrual period of one year
  Determined for each potential participant approached to participate in this study (pre-screened), indicating whether or not the participant was enrolled (underwent blood draw to test for monoclonal gammopathy).

SECONDARY OUTCOMES:
Monoclonal Gammopathy at Screening | From enrollment to availability of lab results, approximately 30 days
  A categorical variable will be determined for each enrolled participant indicating whether or not the participant had monoclonal gammopathy identified on screening blood draw, or if the test results were indeterminate (options: monoclonal gammopathy, no monoclonal gammopathy, unknown/indeterminant test results).
PCD Diagnosis at Screening | From enrollment to completion of diagnostic work up, approximately 90 days
  PCD diagnosis at screening will be determined as a nominal categorical variable indicating the participant's PCD diagnosis at screening. The categorical variable will include the following factor levels: monoclonal gammopathy of undetermined significance (MGUS), smoldering multiple myeloma (SMM), multiple myeloma (MM), AL amyloidosis, other PCD/ lymphoproliferative disorder, monoclonal gammopathy with unknown diagnosis, or no monoclonal gammopathy. Reason for unknown diagnosis may be due to non-definitive results, no results due to lab error, sampling issues, or participant did not get complete diagnostic work up.
PCD Diagnosis During Follow-Up | From enrollment to completion of follow up (10 years)
  PCD diagnosis during follow-up will be determined as a categorical variable for each new PCD diagnosis indicating whether the participant had the type of PCD diagnosed over the course of the follow up period on the study. The types of new PCD diagnosis will include SMM, MM, AL amyloidosis, and other PCD diagnosis, per diagnostic criteria as defined in Appendix A. Date of each new PCD diagnosis will also be captured.
CRAB Criteria at MM Diagnosis | From enrollment to completion of follow up (10 years)
  CRAB criteria at MM diagnosis are defined as a binary variable indicating whether the participant had CRAB criteria at the time of MM diagnosis. CRAB criteria include hypercalcemia, renal insufficiency, anemia, or bone lesions as defined per IMWG. This will be evaluated only in the subjects diagnosed with MM during longitudinal follow-up
Time to MM Diagnosis | From enrollment to completion of follow up (10 years)
  Time to MM diagnosis is defined as the duration of time from MGUS diagnosis (or SMM diagnosis for participants diagnosed with SMM at screening) to diagnosis of MM per IMWG criteria. The date of MM diagnosis is the date of the first assessment that identified MM. If the participant died without a diagnosis of MM, time to MM diagnosis will be calculated at the date of death, with death as a competing risk event. For surviving subjects who do not have documented MM diagnosis, time to MM diagnosis will be censored at the date of the last documented disease evaluation that confirmed no MM diagnosis.
Number of Participants who Interacted with a Community Champion | Baseline
  Interaction with a community champion will be captured for each potential participant as a binary variable indicating whether or not the potential participant interacted with a study-associated community champion prior to enrollment or prior to declining participation. This will be captured via the "Interaction with Community Champion Survey".
Impact of Interaction with a Community Champion | Baseline
  Community champion impact will be reported by each enrolled participant that interacted with a community champion. It will be captured as an ordered categorical variable (5-point Likert scale) indicating the level of impact that the community champion had on the participant's decision to participate in the study. This will be captured via the "Interaction with Community Champion Survey".
Number of MGUS Participants who Participate in Longitudinal Portion of Study | From enrollment to presentation of second (longitudinal) consent, approximately 90 days
  For each participant that is determined to have MGUS at screening, a binary variable will be captured, indicating whether or not the participant consented to be followed longitudinally in the longitudinal portion of the study.
Barriers to Screening Participation | Baseline
  For participants who are approached but do not verbally agree to participation in the study, verbal reason for declining study participation will be reported and captured via a "Barriers to Participation Survey" that includes multi-select discrete options as well as an "Other" reason with free text option.
Barriers to Longitudinal Participation | From enrollment to presentation of second (longitudinal) consent, approximately 90 days
  For participants with monoclonal gammopathy identified during screening but who do not agree to participate in the longitudinal portion of the study, reason for declining longitudinal participation will be reported and captured via a "Barriers to Participation Survey" that includes multi-select discrete options as well as an "Other" with free text option.
Psychological Counseling Referral | From enrollment to completion of diagnostic work up, approximately 90 days.
  For each participant with monoclonal gammopathy identified during screening, a binary variable indicating whether a psychological counseling referral was accepted after learning of positive results.
Light Chain MGUS Diagnosis at Screening | From enrollment to completion of diagnostic work up, approximately 90 days.
  Determined as a binary variable indicating whether the participant had light chain MGUS diagnosis at screening. Three definitions of light chain MGUS (with applicable reference ranges for FLC ratio, involved FLC) will be utilized to evaluate this endpoint: standard IMWG diagnostic criteria [with FLC ranges from Katzmann et al (2002)], iStop MM criteria incorporating age and renal function [Long et al (2025)], and Dana Farber Cancer Institute criteria incorporating race [Bertamini et al (2025)].

CONTACTS AND LOCATIONS:
Overall Officials: Manisha Bhutani, MD, Principal Investigator — Atrium Health Wake Forest Baptist Comprehensive Cancer Center
Locations (1):
- Atrium Health Levine Cancer, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided